CLINICAL TRIAL: NCT06736834
Title: Sensory Evaluation of Chinese Specialty Foods
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Sensory Evaluation
Record Dates: First submitted 2024-12-08; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Dietary Preferences; Sensory Evaluation; Healthy Individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- College students participating in sensory evaluation (Experimental): Youtiao and porridge with different processing time and temperature
  Interventions: Other: Babao Congee and Youtiao(deep-fried dough sticks) with different cooking conditions

INTERVENTIONS:
Other: Babao Congee and Youtiao(deep-fried dough sticks) with different cooking conditions — Babao Congee and deep-fried dough sticks with different cooking conditions

SUMMARY:
This project aims at college student consumers, recruiting a certain number of college student volunteers as sensory evaluators, and requiring them to evaluate samples of Babao Congee and deep-fried dough sticks.

DETAILED DESCRIPTION:
The specific evaluation methods are as follows: the samples are randomly numbered and distributed to college student volunteers. Scale method is used to quantify the appearance score, texture score and taste score of Babao Congee and deep-fried dough sticks. Basic information, general physical conditions and sensory characteristics of Babao Congee and deep-fried dough sticks are collected through questionnaires or interviews.

ELIGIBILITY:
Inclusion Criteria:

* University students at school

Exclusion Criteria:

* Smoking (≥1 cigarette/week);
* heavy alcohol consumption (>224 g/week for men and >168 g/week for women);

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-12-18 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
preference | Each sensory evaluation should be conducted within 2 hours, and for different batches of personnel, the overall time should be completed within one month
  Personnel evaluate and score the color, aroma, taste, and other aspects of food.

IPD SHARING:
Plan to Share IPD: No